CLINICAL TRIAL: NCT03314441
Title: Effects of Regular Practice of Yoga on Subjective and Objective Sleep Quality in Primary Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Chef de Clinique, Centre Hospitalier Universitaire Saint Pierre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE076201733641
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Primary Insomnia
Keywords: yoga; sleep quality; sleep quantity; sleep efficiency; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: 4 yoga lessons with and instructors on a 3 months period. Patients are asked to exercise yoga daily for 5 to 30 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga (Experimental): Patients receiving Yoga lessons for 3 months
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — 4 yoga lessons with and instructors on a 3 months period. Patients are asked to exercise yoga daily for 5 to 30 minutes.

SUMMARY:
The purpose of the study is to assess the effects of regular Viniyoga in patients suffering from primary insomnia.

DETAILED DESCRIPTION:
Insomnia is very prevalent in Europe (14-27%). Cognitive behavioral therapy is the treatment of choice in patients suffering from primary insomnia, allowing to obtain a long term (2 years) sleep quality improvements in 62% of patients. Yoga is another behavioral therapy that have shown benefits in patients suffering from anxiety disorders. Few studies have been focused on yoga benefits in sleep disorders. The purpose of the study is to assess the effects of regular Viniyoga on sleep quality (subjective and objective) in patients suffering from primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

-primary insomnia

Exclusion Criteria:

* shift work,
* associated sleep disorder (sleep apnea, narcolepsy,..)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
total sleep time | 3 months
  total sleep time measured by polysomnography and actigraphy

SECONDARY OUTCOMES:
sleep latency | 3 months
  sleep latency measured by polysomnography and actigraphy
sleep efficiency | 3 months
  sleep efficiency measured by polysomnography and actigraphy
wake after sleep onset | 3 months
  wake after sleep onset measured by polysomnography and actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, PhD, Principal Investigator — CHU St Pierre
Locations (1):
- CHu Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turmel D, Carlier S, Bruyneel AV, Bruyneel M. Tailored individual Yoga practice improves sleep quality, fatigue, anxiety, and depression in chronic insomnia disorder. BMC Psychiatry. 2022 Apr 14;22(1):267. doi: 10.1186/s12888-022-03936-w. PMID 35421962